CLINICAL TRIAL: NCT02672436
Title: A Randomized, Double-Blind, Vehicle-controlled, Parallel, Phase II Study to Evaluate Efficacy and Safety of ENERGI-F703 in Subjects With Diabetic Foot Ulcers
Brief Title: ENERGI-F703 for Diabetic Foot Ulcers Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Energenesis Biomedical Co., Ltd. (Industry)
Collaborators: A2 Healthcare Taiwan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENERGI-F703-01
Record Dates: First submitted 2016-01-27; First posted 2016-02-03 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Foot; Foot Ulcer; Diabetes Mellitus; Wounds
Keywords: Diabetic Foot Ulcer; Diabetes Mellitus; Wound Healing
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Diabetes Mellitus; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ENERGI-F703 (Experimental): ENERGI-F703, topical application, 2 times daily for 12 weeks
  Interventions: Drug: ENERGI-F703
- Placebo (Placebo Comparator): ENERGI-F703 matched vehicle, topical application, 2 times daily for 12 weeks
  Interventions: Drug: ENERGI-F703 matched vehicle

INTERVENTIONS:
Drug: ENERGI-F703 — Standard of care and ENERGI-F703 are applied for treatment of diabetic foot ulcers.
  Arms: ENERGI-F703
Drug: ENERGI-F703 matched vehicle — Standard of care and ENERGI-F703 matched vehicle are applied for treatment of diabetic foot ulcers.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of ENERGI-F703 in subject with diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. With either gender aged at least 20 years old
2. With diagnosed diabetic mellitus (DM), e.g. currently under DM medication treatment or naïve DM subject with duplicated HbA1c over 6.5% and fasting plasma glucose over 126 mg/dL measured at least one week apart before Screening)
3. With at least one cutaneous ulcer on the foot (including ulcers on the lower legs) and not healing for at least 4 weeks. The largest diabetic foot ulcer will be selected as target ulcer. If two or more ulcers have the largest size, the one with worst grade will be selected. If two or more ulcers have the largest size and grade, the one with longest duration will be selected.
4. The target ulcer is classified as grade 1 to 3 ulcer according to Wagner Grading System and with ulcer size of 1 cm2 to 36 cm2 (Grade 3 ulcer subject may enter the study only if after debridement, the abscess of target ulcer is under control at investigator's discretion and osteomyelitis does not present)
5. Diabetic foot ulcers should be free of any necrosis or infection in any soft tissue and bone tissue;
6. Subject has signed the written informed consent form

Exclusion Criteria:

1. With active osteomyelitis
2. With target ulcer size decreased by at least 30% after at least 2 weeks of standard-of-care-only period or any other recorded regular therapy either before Screening visit or after completing Initial Phase
3. With poor nutritional status (albumin < 2g/dl), poor diabetic control (HbA1c > 12%), a leukocyte counts < 2,000/mm3, abnormal liver function (AST, ALT>3 x upper limit of normal range) within 14 days before Screening visit or 28 days before Randomization visit Note: HbA1c: hemoglobin A1c; AST: aspartate aminotransferase; ALT: alanine aminotransferase
4. Requiring treatment with systemic corticosteroids, immunosuppressive or chemotherapeutic agents
5. With known or suspected hypersensitivity to any ingredients of study product and vehicle
6. With coronary heart disease with myocardial infarction, coronary artery bypass graft (CABG), or percutaneous transluminal coronary angioplasty (PTCA) within 3 months prior to study
7. Pregnant or lactating or premenopausal with childbearing potential but not taking reliable contraceptive method(s) during the study period Note: Women with childbearing potential should agree to use a highly effective method of birth control, defined as those, alone or in combination, that result in a low failure rate when used consistently and correctly.
8. With the following conditions:

   1. ankle brachial index (ABI) < 0.4 OR
   2. ABI between 0.4 and 0.6 (inclusive) and not received appropriate treatment for improving venous and arterial insufficiency Note: Subjects with ABI between 0.4 and 0.6 (inclusive) and having received appropriate surgical or endovenous/endovascular therapy for improving venous and arterial insufficiency considered by investigators such as valvuloplasty, angioplasty, or bypass grafting will be eligible to enter the study at investigator's discretion.
9. Enrollment in any investigational drug trial within 4 weeks before entering this study
10. With any condition judged by the investigator that entering the trial may be detrimental to the subject

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
The ulcer closure rate | Week 12
  Defined as the proportion of subjects with complete ulcer closure at the end of treatment period

SECONDARY OUTCOMES:
The accumulated confirmed ulcer closure rate at each of the post-treatment visit | Week 1, 2, 4 ,6 ,8, 10, 12
The ulcer closure time | Week 1, 2, 4, 6, 8, 10, 12
  Defined as the time to complete ulcer closure
Percentage change in ulcer size for each post-treatment visit | Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24
  Calculated as (Ulcer size at post treatment visit - Ulcer size at baseline)/(Ulcer size at baseline)
Adverse event incidence | Week 1, 2, 4, 6, 8, 10, 12, 14, 16, 20, 24

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang JY, Chen CC, Chang SC, Yeh JT, Huang HF, Lin HC, Lin SH, Lin YH, Wei LG, Liu TJ, Hung SY, Yang HM, Chang HH, Wang CH, Tzeng YS, Huang CH, Chou CY, Lin YS, Yang SY, Chen HM, Lin JT, Cheng YF, Young GH, Huang CF, Kuo YC, Dai NT. ENERGI-F703 gel, as a new topical treatment for diabetic foot and leg ulcers: A multicenter, randomized, double-blind, phase II trial. EClinicalMedicine. 2022 Jul 10;51:101497. doi: 10.1016/j.eclinm.2022.101497. eCollection 2022 Sep. PMID 35844773